CLINICAL TRIAL: NCT00752583
Title: Clinical Study in Order to Quantify Solute Removal in Peritoneal Dialysis Versus Haemodialysis
Brief Title: Peritoneal Dialysis Versus Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008/232
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Hemodialysis
Keywords: Chronic renal insufficiency (patients under dialysis)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Peritoneal Dialysis; Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Peritoneal dialysis
  Interventions: Procedure: Peritoneal dialysis
- 2 (Active Comparator): Haemodialysis
  Interventions: Procedure: Haemodialysis

INTERVENTIONS:
Procedure: Peritoneal dialysis — Blood, urine and dialysate sampling
  Arms: 1
Procedure: Haemodialysis — Blood, urine and dialysate sampling
  Arms: 2

SUMMARY:
Study in order to quantify toxin removal during dialysis

ELIGIBILITY:
Inclusion Criteria:

* Substudy 1: includes new starting dialysis patients on peritoneal dialysis PD or haemodialysis HD
* Substudy 2: stabile haemodialysis patients and peritoneal dialysis patients. Patients will be matched for gender, time on dialysis, diabetes, renal function at the start of dialysis.
* Substudy 3: patients on CAPD (continuous ambulant PD) or CCPD (continuous cyclic PD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11-07 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Registration of toxin removal efficiency | After 1 week and after 1, 3, 6, 9, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be